CLINICAL TRIAL: NCT02028702
Title: Alternative Treatments for Menopausal Women: The Efficacy of a Novel Red Clover Treatment on Menopausal Women.
Brief Title: Alternative Treatments for Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Per Bendix Jeppesen, Associate Prof., PhD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Mntl-1877
Record Dates: First submitted 2012-07-12; First posted 2014-01-07 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Menopause; Hot Flushes; Osteoporosis; Dyslipidemia
Keywords: red clover; menopause; bioactive compounds; isoflavones; phytoestrogen
MeSH Terms: conditions — Hot Flashes; Osteoporosis; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red Clover extract (Active Comparator): 150 ml/d Red Clover extract
  Interventions: Dietary Supplement: Red Clover extract
- Placebo (Placebo Comparator): 150 ml/d sweetened and coloured water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — water with color
  Arms: Placebo
Dietary Supplement: Red Clover extract — Red Clover extract containing 80 mg Isoflavones. Dosage: 2 X 75 ml/day
  Other Names: fermentated Red Clover extract
  Arms: Red Clover extract

SUMMARY:
To investigate the reported health benefits (lipid profile, inflammatory factors, cardiovascular status and bone density) of a novel, phytoestrogen rich, Red Clover treatment on women suffering from both menopause related primary (hot flushes, night sweats, sleep disturbance and weight gain) and secondary (osteoporosis, cardiovascular and changes in lipid metabolism) symptoms.

DETAILED DESCRIPTION:
Menopausal symptoms are a common phenomenon causing discomfort to many middle aged women throughout the world. The core symptoms are experienced as hot flushes (HF), night sweats, vaginal dryness and sleep disturbance. Other secondary symptoms are sexual dysfunction, depression, anxiety, memory loss, fatigue, headache, joint pains and weight gain. Moreover there is increased risk of further complications such as osteoporosis, cardiovascular and negative changes in lipid profile associated with the reduction in oestrogen during and post menopause.

Trifolium Pratense or Red Clover (RC) has arisen as a popular source for women experiencing HF because it contains a variety of phytoestrogen's, namely isoflavones, lignans and coumestans. Phytoestrogens are shown to have positive effects on menopausal disorders such as breast cancer, cardiovascular risk factors, osteoporosis and have been shown to exert non-hormonal antioxidant effects. Additionally these isoflavones appear to reduce bone resorbtion, help maintain bone mineral density and improve lipid profile (reducing LDL: HDL, lipoprotein A, total cholesterol and may also reduce triglycerides).

RC is particularly high in estrogenic isoflavones biochanin A, formononetin and to a lesser degree genestein and diadzein, although the two former are precursors to genestein and diadzein. Asian populations with a high intake of soy (rich in genestein and diadzein) have long shown a lower reported incidence of the symptoms of menopause.

The study will be carried out as a 3-month parallel randomized control intervention study, consisting of 61 menopausal women. During summer 2012, 61 participants will be randomised into 2 groups (~30-31 in each group). The two groups are as follows:

1. Menopausal women receiving RC treatment - 150ml/d Red Clover (80mg/d of isoflavones as aglycone)
2. Menopausal women receiving placebo - 150ml placebo

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-65 years
* Experiencing daily hot flushes
* Body Mass Index (BMI) between 20-40
* Irregular menstrual bleeding
* FSH levels above the normal range

Exclusion Criteria:

* Simultaneous participation in other clinical trials within the last 3 months
* Severe cardiovascular, psychiatric, neurological, and/or kidney disease.
* Alcohol or drug abuse and acute illness.
* Blood pressure > 160/110
* Pregnant and lactating women

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary Menopause-related symptoms | 3 months
  To examine the extent to which red clover extract can reduce the frequency and intensity of hot flashes, sleep disturbances and flush related sweats.

CONTACTS AND LOCATIONS:
Overall Officials: Per B Jeppesen, Prof, Principal Investigator — Aarhus University Hospital
Locations (1):
- Center for Clinical Research, Hospital Vendsyssel, Hjørring, North Denmark, Denmark

REFERENCES:
- [Derived] Lambert MNT, Thorup AC, Hansen ESS, Jeppesen PB. Combined Red Clover isoflavones and probiotics potently reduce menopausal vasomotor symptoms. PLoS One. 2017 Jun 7;12(6):e0176590. doi: 10.1371/journal.pone.0176590. eCollection 2017. PMID 28591133